CLINICAL TRIAL: NCT02891278
Title: The Clinical Application of Tumor Reversion: A Phase I Study of Sertraline (Zoloft) in Combination With Timed-sequential Cytosine Arabinoside (Ara-C) in Adults With Relapsed and Refractory Acute Myeloid Leukemia (AML)
Brief Title: Sertraline and Cytosine Arabinoside in Adults With Relapsed and Refractory AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Joseph Jurcic, Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ8444; 6474-15 (Other Grant/Funding Number: Leukemia and Lymphoma Society)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Leukemia; Sertraline; Cytosine Arabinoside; Relapsed AML; Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Sertraline; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sertraline with cytosine arabinoside (Experimental): All subjects will receive the following:
  Induction phase
  * Sertraline, twice daily at one of the pre-defined dose levels
  * Cytosine arabinoside, on days 1 and 10
  Consolidation phase
  Patients who achieve complete remission (CR) or complete remission with incomplete count recovery (CRi) and are eligible for allogeneic stem cell transplantation will receive one of the following:
  * Allogeneic SCT and off study
  * Repeat cycle of oral sertraline and cytosine arabinoside IV infusion
  * Maintenance phase with sertraline for cycles of 28 days in length
  Interventions: Drug: Sertraline; Drug: Cytosine arabinoside; Procedure: allogeneic stem cell transplantation

INTERVENTIONS:
Drug: Sertraline — Sertraline is a selective serotonin reuptake inhibitor (SSRI) that is FDA approved to treat major depressive disorder, obsessive-compulsive disorder, panic disorder, post-traumatic stress disorder, premenstrual dysphoric disorder, and social anxiety disorder.
  Sertraline will be administered orally twice a day starting on day -3. Sertraline will be administered at one of 4 pre-defined dose levels in the following dose-escalation: 50 mg daily, 50 mg twice a day, 50 mg every morning (QAM) and 100 mg every evening (QPM), 100 mg twice a day. 100 mg QAM and 150 mg QPM.
  Other Names: Zoloft
Drug: Cytosine arabinoside — Cytarabine is a cytotoxic chemotherapy approved for use in acute myeloid leukemia, acute lymphoblastic leukemia, and chronic myelogenous leukemia. It is also approved to prevent and treat meningeal leukemia. Cytarabine kills cells in S-phase through inhibition of DNA polymerase, as well as by halting DNA synthesis after its incorporation into DNA.
  Cytosine arabinoside (Ara-C) will be administered as a 72 hour intravenous continuous infusion (IVCI) beginning Day 1 of therapy and again beginning Day 10 of therapy. The total dose of ara-C for each 72 hour period is 2 gm/m2 (0.667 gm/m2/24 hours).
  Other Names: ara-C; Cytarabine
Procedure: allogeneic stem cell transplantation — Allogeneic stem cell transplantation involves transferring the stem cells from a healthy person (the donor) to a patient after high-intensity chemotherapy or radiation.
  Other Names: allogeneic SCT

SUMMARY:
This is a Phase I study with the goals of determining the feasibility, safety, and toxicity of administering sertraline in combination with timed-sequential cytosine arabinoside (ara-C) in adults with relapsed and refractory acute myeloid leukemia (AML).

Primary objective:

* To define the maximum tolerated dose (MTD) and Recommended Phase II Dose (RP2D) of sertraline administered in combination with timed-sequential cytosine arabinoside in adult patients with relapsed and refractory acute myeloid leukemia.
* To evaluate the safety and tolerability of sertraline given in combination with timed-sequential cytosine arabinoside in adult patients with relapsed and refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
Relapsed and refractory acute myeloid leukemias are characterized by net drug resistance. At the root of this drug resistance is an enhanced survival that relates to intrinsic cell cycle dysregulation and aberrations in the overall process of the repair of DNA damage. These malignancies represent a continuing therapeutic challenge, since currently no "standard treatments" for these diseases exist. Approximately 30% of adults with newly diagnosed AML are primary refractory to chemotherapy and at least 50% of those who achieve remission will relapse. For patients with relapsed or refractory AML, the expected CR/CRi rates with traditional multi-agent chemotherapies range from < 10% for primary refractory AML to 25-30% for relapsed AML and cure rates < 20%, even with allogeneic stem cell transplantation. Thus, novel treatment approaches are needed.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed diagnoses of relapsed AML: Patients with AML that have relapsed at least once or are primary induction failure will be eligible
* Age ≥ 18 and ≤ 70 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2
* ≥ 2 weeks off cytotoxic chemotherapy
* ≥ 2 weeks off radiation therapy
* Off biologic therapies including hematopoietic growth factors ≥ 1 week
* If using tyrosine kinase inhibitors (TKIs)/src inhibitors, other non-cytotoxics, or leukopheresis for blast count control, the patient must be off these therapies for > 24 hrs before starting sertraline. Hydroxyurea will be allowed with sertraline but should be stopped ≥24 hours before starting cytarabine.
* Adequate organ function as defined below:

  * Renal function: Serum creatinine <2.0 mg/dL or creatinine clearance ≥ 50 mL/minute
  * Hepatic function: aspartate aminotransferase (AST), alanine aminotransferase (ALT) and Alkaline Phosphatase ≤ 5x Upper Limit normal (ULN), bilirubin ≤ 2.0 mg/dl, unless due to Gilbert's, hemolysis or leukemic infiltration
  * Left Ventricular Ejection Fraction ≥ 45% by multigated acquisition (MUGA) scan or Echocardiogram
* Patients who have undergone stem cell transplantation (SCT), autologous or allogeneic, are eligible provided that they are ≥ 8 weeks from stem cell infusion, have no active graft versus host disease (GVHD), are off immune suppression for at least 2 weeks, and do not have a history of veno-occlusive disease (VOD)
* Female patients of childbearing age must have negative pregnancy test and women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 30 days after study participation
* Patients must be able to give informed consent

Exclusion Criteria:

* Concomitant chemotherapy, radiation therapy, or immunotherapy
* Patients who are receiving any other investigational agents concurrently
* Hyperleukocytosis with ≥ 30,000 blasts/microliter (uL). If using tyrosine kinase/src inhibitors (FLT-3 inhibitors), other non-cytotoxics, or leukopheresis for blast count control, the patient must be off these therapies for ≥ 24 hours prior to beginning sertraline. If using hydroxyurea for blast count control, this may be continued until up to 24 hours before starting cytarabine
* Acute Progranulocytic Leukemia (APL)
* Active central nervous system (CNS) leukemia
* Active, uncontrolled infection. Patients with infection under active treatment and controlled with antibiotics are eligible
* Presence of other life-threatening illness
* Patients with mental deficits and/or psychiatric history that preclude them from giving informed consent or from following protocol
* Pregnant women are excluded from this study due to potential teratogenic and/or abortifacient effect of this combination chemotherapy. Nursing mother should stop breastfeeding to be eligible due to potential risk for adverse events in nursing infant
* Subjects with the following cardiac risk factors must be excluded: transmural myocardial infarction (MI) within prior 6 months, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack (TIA) or seizure disorder within 6 months prior to study drug administration. In addition, patients with New York Heart Association (NYHA) class III or IV heart failure will be excluded
* Patients requiring treatment with other anti-depressive medications including the selective and non-selective monoamine oxidase (MAO) inhibitors (including linezolid), 5-hydroxytryptamine (5-HT) receptor agonists (triptans), tryptophan or antidopaminergic agents (anti-psychotics, metoclopramide, promethazine, haloperidol)
* Patients requiring prolonged treatment with fluconazole, voriconazole, or posaconazole. Use of isavuconazonium sulfate, liposomal amphotericin, are echinocandins are permitted
* Prior treatment with clofarabine within 6 months or history of clofarabine-induced liver dysfunction
* History of hypersensitivity to sertraline
* Patients taking sertraline at the time of study entry will not be eligible for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of sertraline administered in combination with timed-sequential cytosine arabinoside | Up to 24 months
  Standard 3+3 dose-escalation design will be used to determine the MTD. The MTD will be determined as the highest dose level where 1/6 patients experience dose-limiting toxicity (DLT). Three patients will be treated at a given dose level combination and observed for at least 4 weeks to assess toxicity. Doses will not be escalated in any individual patient.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lee, MD, Principal Investigator — Columbia University; Joseph Jurcic, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: No